CLINICAL TRIAL: NCT01266902
Title: An Open-label Trial With TMC278 25 mg q.d. in Combination With a Background Regimen Containing 2 N(t)RTI's in HIV-1 Infected Subjects Who Participated in TMC278 Clinical Trials and Were Still Benefitting From Treatment With TMC278
Brief Title: A Trial With TMC278-TIDP6-C222 for Continued TMC278 Access in Patients Infected With Human Immunodeficiency Virus-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017434; TMC278-TiDP6-C222 (Other: Janssen R&D Ireland); 2010-021209-18 (EudraCT Number)
Expanded Access: NCT03847376 (Approved for marketing)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 Infection; HIV-1; HIV; TMC278-TiDP6-C222; TMC278-C222; TMC278; Rilpivirine
MeSH Terms: interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Rilpivirine (Experimental): Rilpivirine 25 mg once daily
  Interventions: Drug: Rilpivirine

INTERVENTIONS:
Drug: Rilpivirine — 25 mg once daily

SUMMARY:
The purpose of the study is to provide continued access to TMC278 in HIV-1 infected patients who were randomized and treated with TMC278 in the Phase IIb or Phase III trials.

DETAILED DESCRIPTION:
This is a Phase III, open-label (all people know the identity of the drug), multicenter, roll-over trial to provide continued access to TMC278 to HIV-1 infected patients who were randomized (the study drug is assigned by chance) and treated with TMC278 in the Phase IIb (TMC278-C204 [C204]) or Phase III trials (i.e., TMC278-TiDP6-C209 [C209] or TMC278-TiDP6-C215 [C215]) and who continue to benefit from their antiretroviral treatment, according to the investigator. In addition, information on the long-term safety and tolerability, including resistance data in case of virologic failures, of oral doses of TMC278 25 mg once daily (q.d.) in combination with a background regimen containing 2 N(t)RTIs will be collected. Available efficacy data will also be collected. Approximately 750 HIV-1 infected individuals are expected to participate in this trial. The duration of participation in the study for an individual participant will be 2 to 3 years. The final/withdrawal visit of the Phase IIb or Phase III trials will be the first visit of this trial. Safety and tolerability will be evaluated throughout the trial. Visits and assessments performed should be based on the local, generally accepted standard of care, with visits occurring at least every 6 months. Oral tablets of TMC278 25 mg once daily (q.d.) should be administered together with a meal.

ELIGIBILITY:
Inclusion Criteria:

* Patients are HIV-1 infected and were previously randomized to receive TMC278 in a TMC278 clinical trial and completed the protocol-defined treatment period.
* Patients continue to benefit from treatment with TMC278 in the opinion of the investigator.
* Patient can comply with the current protocol requirements.
* The patient's general medical condition, in the investigator's opinion, does not interfere with participation in the trial.

Exclusion Criteria:

* Use of disallowed concomitant therapy.
* Females of childbearing potential who are pregnant, or without the use of effective birth control methods, or not willing to continue practicing these birth control methods during the trial and for at least 1 month after the end of the trial (or last intake of TMC278).
* Non-vasectomized heterosexually active male patients without the use of effective birth control methods or not willing to continue practicing these birth control methods during the trial and for at least 1 month after the end of the trial (or after last intake of TMC278).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (98):
- United States (29):
  - Beverly Hills, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Sacramento, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Albany, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Longview, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Argentina (5):
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Córdoba
  - Guernica
  - Rosario
- Australia (5):
  - Darlinghurst
  - Melbourne
  - Perth
  - Surry Hills
  - Victoria
- Vienna, Austria
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
- Canada (6):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Montreal
- Santiago, Chile
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai
- Denmark (3):
  - Copenhagen
  - Hvidovre
  - Odense
- France (5):
  - Clamart
  - Lyon
  - Nantes
  - Paris
  - Tourcoing
- Germany (6):
  - Berlin
  - Cologne
  - Essen
  - Frankfurt
  - Hamburg
  - Hanover
- Rotterdam, Netherlands
- San Juan, Puerto Rico
- Romania (2):
  - Bucharest
  - Iași
- Russia (7):
  - Kazan'
  - Krasnodar
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Volgograd
  - Voronezh
- South Africa (7):
  - Bloemfontein
  - Dundee
  - Durban
  - Johannesburg
  - Johannesburg Gauteng
  - Pretoria
  - Westdene Johannesburg Gauteng
- Spain (4):
  - Alicante
  - Barcelona
  - Elche
  - Madrid
- Stockholm, Sweden
- Kaohsiung County, Taiwan
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- United Kingdom (3):
  - Brighton
  - London
  - Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total of 482 participants were treated and 437 discontinued at data cut-off date (8 February 2018) because they switched to commercially available rilpivirine (RPV) (371 participants), as planned per protocol. Only 6 of the 482 participants discontinued as they reached a virologic endpoint. At last contact date of last participant under Protocol Amendment 3 (28 February 2020), out of 45 participants 37 switched to commercially available RPV and 6 were lost to follow-up.
Groups:
- Rilpivirine (RPV) (TMC278-C204 [C204]): Participants who rolled over from trial C204 (NCT00110305) continued to receive RPV 25 milligrams (mg) once daily (qd) in combination with an investigator-selected background regimen consisting of 2 nucleos(t)ide reverse transcriptase inhibitors (N[t]RTI)s starting Day 1.
- RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]): Participants who rolled over from trial C209 (NCT00540449) and C215 (NCT00543725) continued to receive RPV 25 mg qd in combination with an investigator-selected background regimen consisting of 2 N(t)RTIs starting Day 1. In trial C209, the background regimen was fixed to tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) and in trial C215, the background regimen was selected by the investigator and contained either abacavir (ABC)/lamivudine (3TC), zidovudine (AZT)/3TC, or TDF/FTC.
- RPV 25 mg (After Protocol Amendment 3): All Participants who were continued under a simplified study setting with only a minimum of study-related activities, as per Protocol Amendment 3 continued to receive RPV 25 mg and followed up for safety.
Period: Period 1 (Main Study)
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]) | RPV 25 mg (After Protocol Amendment 3)
Started | 119 | 363 | 0
Completed | 89 | 282 | 0
Not Completed | 30 | 81 | 0
Not completed — Investigator's decision/Participant's decision | 2 | 3 | 0
Not completed — Lost to Follow-up | 5 | 12 | 0
Not completed — Lack of Efficacy | 4 | 2 | 0
Not completed — Adverse Event | 3 | 11 | 0
Not completed — Withdrawal by Subject | 2 | 12 | 0
Not completed — Subject non-compliant | 3 | 7 | 0
Not completed — Continued RPV treatment | 11 | 34 | 0
Period: Period 2 (After Protocol Amendment 3)
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]) | RPV 25 mg (After Protocol Amendment 3)
Started | 0 | 0 | 45
Completed | 0 | 0 | 37
Not Completed | 0 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]) | Total
Number analyzed (Participants) | 119 | 363 | 482
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8.18) | 39.9 (9.09) | 40.4 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 84 | 125
  Male | 78 | 279 | 357
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 43 | 58 | 101
  Black or African American | 17 | 64 | 81
  Other | 9 | 0 | 9
  White | 50 | 237 | 287
Region of Enrollment [Number; unit: participants]
  ARGENTINA | 19 | 16 | 35
  AUSTRALIA | 0 | 11 | 11
  AUSTRIA | 2 | 6 | 8
  BELGIUM | 0 | 13 | 13
  CANADA | 0 | 21 | 21
  CHILE | 0 | 12 | 12
  CHINA | 8 | 18 | 26
  DENMARK | 0 | 5 | 5
  FRANCE | 5 | 15 | 20
  GERMANY | 3 | 24 | 27
  ITALY | 0 | 10 | 10
  NETHERLANDS | 0 | 3 | 3
  PUERTO RICO | 7 | 0 | 7
  ROMANIA | 0 | 4 | 4
  RUSSIAN FEDERATION | 11 | 27 | 38
  SOUTH AFRICA | 13 | 35 | 48
  SPAIN | 0 | 14 | 14
  SWEDEN | 0 | 3 | 3
  TAIWAN | 0 | 2 | 2
  THAILAND | 34 | 31 | 65
  UNITED KINGDOM | 8 | 17 | 25
  UNITED STATES | 9 | 76 | 85

OUTCOME MEASURES:

1. Secondary Outcome: Time to Virologic Rebound
Description: Time to virologic rebound was time to (first) human immunodeficiency virus type1 (HIV-1) ribonucleic acid (RNA) greater than or equal to (>=) 50 or >=200 copies/milliliter (copies/mL). The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Up to Week 360
Population: The ITT population included all participants who have taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimens.
Measure: Mean (Standard Error); unit: days
Groups:
- Rilpivirine (RPV) (TMC278-C204 [C204]): Participants that rolled over from trial C204 (NCT00110305) continued to receive RPV 25 mg qd in combination with a background regimen consisting of 2 N(t)RTIs starting Day 1.
- RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]): Participants that rolled over from trial C209 (NCT00540449) and C215 (NCT00543725) continued to receive RPV 25 mg qd in combination with a background regimen consisting of 2 N(t)RTIs starting Day 1. In trial C209, the background regimen was fixed to TDF/FTC and in trial C215, the background regimen was selected by the investigator and contained either ABC/3TC, AZT/3TC, or TDF/FTC.
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
days
  >= 50 copies/mL | 1670.6 (51.32) | 1939.3 (52.43)
  >= 200 copies/mL | 1901.3 (47.19) | 1877.3 (25.93)

2. Secondary Outcome: Time To Treatment Failure
Description: Time to treatment failure was defined as time to virologic rebound (time to first HIV-1 RNA >= 50 or >= 200 copies/mL) or discontinuation for reason other than RPV having become commercially available in the participating country, whichever came first, calculated as the time (in days) from baseline until treatment failure. The mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Up to Week 360
Population: The ITT population included all participants who have taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen.
Measure: Mean (Standard Error); unit: days
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
days
  >= 50 copies/mL | 1795.7 (70.03) | 1694.1 (59.42)
  >= 200 copies/mL | 1868.7 (63.29) | 1637.5 (42.42)

3. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Count for Observed Case Approach Until Week 336
Description: The immunologic assessment was determined by change from baseline in CD4+ cell count for observed case approach.
Time Frame: Baseline up to weeks 96, 192, 288, 336
Population: The ITT population included all participants who have taken at least 1 dose of RPV, regardless of their compliance with the protocol and adherence to the dosing regimen. Here 'number of participants analyzed' signifies number of participants analyzed in this outcome measure. Here 'number analyzed' included all participants evaluable at specified timepoint categories.
Measure: Mean (Standard Error); unit: cells/microliter (cells/mcL)
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
cells/microliter (cells/mcL)
  Week 96: number analyzed (Participants) | 74 | 149
  Week 96 | 72.63 (20.581) | 55.91 (13.425)
  Week 192: number analyzed (Participants) | 68 | 100
  Week 192 | 148.76 (24.111) | 132.73 (21.989)
  Week 288: number analyzed (Participants) | 45 | 89
  Week 288 | 122.29 (29.628) | 101.50 (24.108)
  Week 336: number analyzed (Participants) | 12 | 30
  Week 336 | 161.73 (39.851) | 76.49 (40.484)

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count for Non-Completer Equals Failure (NC=F) Approach Until Week 336
Description: Change from baseline in CD4+ cell count were reported for NC=F approach (participants who discontinued because RPV became commercially available or could be accessed through another source or because the participants switched to other local [RPV-based] treatment options or local standard of care, were censored at that time; other participants after discontinuation had their CD4+ values imputed with baseline value. Intermittently missing values were imputed with a last observation carried-forward approach).
Time Frame: Baseline up to weeks 96, 192, 288, 336
Population: as for outcome 3
Measure: Mean (Standard Error); unit: cells/mcL
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
cells/mcL
  Week 96: number analyzed (Participants) | 79 | 196
  Week 96 | 69.76 (19.372) | 42.19 (11.525)
  Week 192: number analyzed (Participants) | 77 | 153
  Week 192 | 133.56 (21.906) | 91.69 (15.563)
  Week 288: number analyzed (Participants) | 61 | 134
  Week 288 | 92.12 (22.809) | 63.33 (17.132)
  Week 336: number analyzed (Participants) | 27 | 86
  Week 336 | 70.69 (23.558) | 49.24 (16.688)

5. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
Participants | 9 | 14

6. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Time Frame: Up to 7 years
Population: The intent-to-treat (ITT) population included all participants who have taken at least 1 dose of rilpivirine (RPV), regardless of their compliance with the protocol and adherence to the dosing regimens.
Measure: Number; unit: Participants
Groups:
- Rilpivirine (RPV) (TMC278-C204 [C204]): Participants that rolled over from trial C204 (NCT00110305) continued to receive RPV 25 milligrams (mg) once daily (qd) in combination with a background regimen consisting of 2 nucleos(t)ide reverse transcriptase inhibitors (N[t]RTI)s starting Day 1.
- RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]): Participants that rolled over from trial C209 (NCT00540449) and C215 (NCT00543725) continued to receive RPV 25 mg qd in combination with a background regimen consisting of 2 N(t)RTIs starting Day 1. In trial C209, the background regimen was fixed to tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC) and in trial C215, the background regimen was selected by the investigator and contained either abacavir (ABC)/lamivudine (3TC), zidovudine (AZT)/3TC, or TDF/FTC.
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
Participants | 32 | 70

7. Primary Outcome: Number of Participants With Grade 3/4 Events of Rash Irrespective of Causality
Description: Number of participants with grade 3/4 events of rash irrespective of causality were assessed. A grade 3 rash defined as diffuse macular, maculopapular or morbilliform rash with vesicles or limited number of bullae or; rash with superficial ulcerations of mucous membranes limited to 1 anatomical site or; rash with at least one of the following: elevations in aspartate aminotransferase (AST)/alanine aminotransferase (ALT) more than 2*baseline value and at least 5 times upper limit of normal; fever greater than (>) 38 degree celsius or 100 degree fahrenheit; eosinophils > 1000/millimeter (mm)^3; serum sickness-like reaction. A grade 4 rash defined as the following: extensive or generalized bullous lesions or; Stevens-Johnsons Syndrome (SJS) or ulceration of mucous membrane involving 2 or more distinct mucosal sites or toxic epidermal necrolysis.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With AEs Related to Rilpivirine (RPV)
Description: Number of participants with AEs related to RPV were assessed. An AE can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Time Frame: Up to 7 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
Number analyzed (Participants) | 119 | 363
Participants | 7 | 16

ADVERSE EVENTS:
Time Frame: Up to 7 years
Description: Safety analysis included all participants who have taken at least 1 dose of rilpivirine (RPV), regardless of their compliance with the protocol and adherence to the dosing regimen.
Arm/Group | Rilpivirine (RPV) (TMC278-C204 [C204]) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215])
All-Cause Mortality (participants affected / at risk) | 0/119 | 2/363
Serious Adverse Events (participants affected / at risk) | 9/119 | 16/363
Other Adverse Events (participants affected / at risk) | 25/119 | 61/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rilpivirine (RPV) (TMC278-C204 [C204]) (N=119) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]) (N=363)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac hypertrophy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rilpivirine (RPV) (TMC278-C204 [C204]) (N=119) | RPV (TMC278-TiDP6-C209 [C209] and TMC278-TiDP6-C215 [C215]) (N=363)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Feeling hot (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Body tinea (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Chlamydial infection (Infections and infestations) | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0
Eye infection toxoplasmal (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 2
Hordeolum (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Latent tuberculosis (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Syphilis (Infections and infestations) | 2 | 2
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
Blood lactic acid increased (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 3
Liver function test abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cluster headache (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 4
Paraesthesia (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 7
Abnormal dreams (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Facial wasting (Skin and subcutaneous tissue disorders) | 2 | 0
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Not all Adverse Events (AEs) were collected; AEs considered related to rilpivirine (RPV), leading to discontinuations, serious adverse events (SAEs), or grade 3/4 events of rash regardless of causality were collected; discontinuation rate was greater than (>) 90 percent which makes interpretation of results difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT01266902/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/02/NCT01266902/SAP_001.pdf